CLINICAL TRIAL: NCT00790634
Title: Characterizing Mechanisms of Fronto-Subcortical Dysfunction: A Comparison Between Parkinson's Disease and Obsessive-Compulsive Disorder
Brief Title: Mechanisms of Fronto-Subcortical Dysfunction: Comparing PD and OCD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: University of Haifa (Other); Israel Science Foundation (Other)
Responsible Party: Dr. Sharon Hassin, principal investigator, Sheba Medical Center
Other Study IDs: SHEBA-08-5473-SH-CTIL
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Parkinson's Disease; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Parkinson Disease; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Parkinson's Disease: Patients with idiopathic Parkinson's disease
- Obsessive-compulsive disorder: Individuals with a diagnosis of obsessive-compulsive disorder
- OCD controls: Healthy controls, matched in age and number to obsessive-compulsive group
- PD controls: Healthy controls, matched in age and number to Parkinson's disease group

SUMMARY:
The purpose of this study is to characterize and compare irregularities in dopaminergic function in fronto-subcortical circuits, between Parkinson's Disease patients (ON and OFF medication) and patients with obsessive-compulsive disorder, by examining performance on cognitive tasks involving cognitive flexibility, decision-making, and attentional bias.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD or
* OCD
* for control group - age-matched to study groups

Exclusion Criteria:

* psychotic symptoms (past or present)
* head injury with loss of consciousness
* other neurological conditions (excepting PD in PD group)
* for OCD group - use of dopaminergic medications

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: private and hospital-based clinics, healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)